CLINICAL TRIAL: NCT05478551
Title: Randomized Controlled Trial Examining the Efficacy of Botulinum Toxin in Biopsy Scar Minimization
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, David M. Ozog, Department Chair, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15432
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Scar; Hypertrophic Scar
Keywords: botulinum toxin; scar prevention; scar formation
MeSH Terms: conditions — Cicatrix; Cicatrix, Hypertrophic | interventions — Botulinum Toxins; abobotulinumtoxinA; Saline Solution

STUDY DESIGN:
Intervention Model Description: We will be conducting a split-scar study/study involving two biopsy sites in a singular patient, allowing them to serve as their own control.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The injector, assessor, patient, and outcome assessor will be blinded to the treatment side and placebo side of injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Botulinum toxin (Experimental): Biopsy site receiving botulinum toxin
  Following the biopsy closures, one of two biopsy sites (left or right) will be selected to receive 30u (0.3cc) of botulinum toxin injected into the suture line at a depth of PPD bleb.
  The treatment for each wound site will be randomized (left versus right) and blinded but consistent throughout dosing.
  Interventions: Drug: Botulinum Toxin
- Placebo (Placebo Comparator): Placebo Comparator: Biopsy site receiving placebo
  Following the biopsy closures, the other biopsy site will receive 30u (0.3cc) of bacteriostatic normal saline injected into the suture line at a depth of PPD bleb.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Botulinum Toxin — We will be comparing botulinum toxin following the biopsies to placebo injection. We will then compare photos of each biopsy site at set intervals following the procedure.
  Other Names: Dysport; BTXa; abobotulinumtoxinA
  Arms: Botulinum toxin
Drug: Normal saline — Normal saline will serve as the placebo control on the contralateral side of the back.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The proposed study seeks to evaluate the scar reduction capacity of BTA on excision/biopsy wounds compared to the control (normal saline) in a double-blinded randomized control trial. It will expand upon previous studies that have already demonstrated the safety and good tolerance profile of BTA. We will be conducting a split-scar study/study involving two biopsy sites in a singular patient, allowing them to serve as their own control. In keeping with the results from previously conducted studies, we hypothesize that the wounds treated with BTA will have significantly less evidence of scar formation than those sites treated with normal saline.

DETAILED DESCRIPTION:
The process of scar formation is denoted by three stages: inflammatory, proliferative, and remodeling. The former phase is characterized by the activation of the extrinsic clotting pathway and subsequent materialization of a fibrin plug, after which neutrophils facilitate the degradation of pathogens and secretion of signaling molecules that commence the proliferative phase. The fibrin plug is then replaced by granulation tissue comprised of macrophages, fibroblast, and endothelial cells in the proliferative phase. Through the release several growth factors, existing macrophages induce laying down of type III collagen by fibroblasts, and keratinocytes work in tandem to approximate wound edges. Lastly, during the remodeling phase, cellular apoptosis causes granulation tissue formation to subside, type III collagen is replaced by a more durable collagen type I, and myofibroblasts help to condense the scar size.1,2

While scarring in its non-pathological forms is an innate and appropriate bodily response to cutaneous injury, scar development and persistence can have negative physical and psychological implications, including decreased range of motion secondary to contracture, disfigurement, and impaired quality of life.1,3-5 Thus, for medical and cosmetic purposes alike, curtailing scar formation is important aspect of patient management, and treatment aimed at both prevention and resolution is an evolving subject in the medical discourse. Credence has been given to the use of botulinum toxin A (BTA) in scar minimization, a more novel therapy, and has proved efficacious in several studies including those examining BTA in the treatment of keloids and hypertrophic scars, mammoplasty and abdominoplasty surgery scars, and post-operative scars generally.6-9 The suggested mechanisms for this phenomenon involve inhibition of pre-synaptic acetylcholine channels that lead to muscle paralysis and relaxation of perpendicular wound tension; this particular mechanism is likewise theorized to mitigate collagen overproduction. Another hypothesis for explaining the ability of BTA to reduce scar appearance is the direct modulation of fibroblast activity.6

ELIGIBILITY:
Inclusion Criteria:

* Healthy Individuals age 18 and older
* Able to understand the requirements of the study and its associated risks
* Able to complete and sign a consent form

Exclusion Criteria:

* Allergy to botulinum toxin
* Currently pregnant or breastfeeding
* Myasthenia gravis
* Previous injection of botulinum toxin in the specified treatment areas within 6 months prior to enrollment
* Unable to follow up 6 months after biopsy procedure
* Refusal to participate in the trial
* History of keloid or hypertrophic scars
* Eaton-Lambert Syndrome
* Amyopathic Lateral Sclerosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 3 months
  Modified Patient and Observer Scar Assessment Scale v2.0 (POSAS)
Primary Outcome Measure | 6 months
  Modified Patient and Observer Scar Assessment Scale v2.0 (POSAS)

CONTACTS AND LOCATIONS:
Overall Officials: David Ozog, MD, Principal Investigator — Henry Ford Health Systems
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There will be a publication based on the results of the study. We will not be sharing individual participant data outside of our institution and all data collected will be kept on a secured drive within the Henry Ford Health System.

REFERENCES:
- [Result] Tziotzios C, Profyris C, Sterling J. Cutaneous scarring: Pathophysiology, molecular mechanisms, and scar reduction therapeutics Part II. Strategies to reduce scar formation after dermatologic procedures. J Am Acad Dermatol. 2012 Jan;66(1):13-24; quiz 25-6. doi: 10.1016/j.jaad.2011.08.035. PMID 22177632
- [Result] Kasyanju Carrero LM, Ma WW, Liu HF, Yin XF, Zhou BR. Botulinum toxin type A for the treatment and prevention of hypertrophic scars and keloids: Updated review. J Cosmet Dermatol. 2019 Feb;18(1):10-15. doi: 10.1111/jocd.12828. Epub 2018 Dec 12. PMID 30548742
- [Result] Oosterwijk AM, Mouton LJ, Schouten H, Disseldorp LM, van der Schans CP, Nieuwenhuis MK. Prevalence of scar contractures after burn: A systematic review. Burns. 2017 Feb;43(1):41-49. doi: 10.1016/j.burns.2016.08.002. Epub 2016 Sep 14. PMID 27639820
- [Result] Oh H, Boo S. Assessment of burn-specific health-related quality of life and patient scar status following burn. Burns. 2017 Nov;43(7):1479-1485. doi: 10.1016/j.burns.2017.03.023. Epub 2017 May 21. PMID 28539239
- [Result] Ziolkowski N, Kitto SC, Jeong D, Zuccaro J, Adams-Webber T, Miroshnychenko A, Fish JS. Psychosocial and quality of life impact of scars in the surgical, traumatic and burn populations: a scoping review protocol. BMJ Open. 2019 Jun 3;9(6):e021289. doi: 10.1136/bmjopen-2017-021289. PMID 31164358
- [Result] Abedini R, Mehdizade Rayeni N, Haddady Abianeh S, Rahmati J, Teymourpour A, Nasimi M. Botulinum Toxin Type A Injection for Mammoplasty and Abdominoplasty Scar Management: A Split-Scar Double-Blinded Randomized Controlled Study. Aesthetic Plast Surg. 2020 Dec;44(6):2270-2276. doi: 10.1007/s00266-020-01916-7. Epub 2020 Aug 19. PMID 32813130
- [Result] Yang W, Li G. The Safety and efficacy of botulinum toxin type A injection for postoperative scar prevention: A systematic review and meta-analysis. J Cosmet Dermatol. 2020 Apr;19(4):799-808. doi: 10.1111/jocd.13139. Epub 2019 Sep 12. PMID 31513335
- [Result] Guo X, Song G, Zhang D, Jin X. Efficacy of Botulinum Toxin Type A in Improving Scar Quality and Wound Healing: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Aesthet Surg J. 2020 Apr 14;40(5):NP273-NP285. doi: 10.1093/asj/sjz165. PMID 31155638